CLINICAL TRIAL: NCT02846220
Title: Overcoming Immunity to Change: A Feasibility Study of a New Method to Promote Medication Adherence Among Older Adults With Hypertension
Brief Title: Promoting Medication Adherence Among Older Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: Minds at Work (Unknown); Ohio State University (Other)
Responsible Party: Principal Investigator, Marie Krousel-Wood, Professor, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 735133
Record Dates: First submitted 2016-05-24; First posted 2016-07-27 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Hypertension
Keywords: Medication Adherence; Middle Aged 45-64; Aged 65-79; Aged, 80 and over
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health coaching (Experimental): Two-hour in-person group counseling session led by health coach, involving development of personalized immunity maps that lay out adherence goal, behaviors that distract from goal, hidden motives that compete with achieving goal, and underlying assumptions
  Eight 50-minute individual telephone counseling sessions every three weeks with a health coach, focusing on uncovering hidden motives and challenging assumptions with the goal of overturning nonadherence mindsets
  Interventions: Behavioral: Overcoming Immunity to Change health coaching
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Overcoming Immunity to Change health coaching
  Arms: Health coaching

SUMMARY:
Over 70% of US adults 65 or older are diagnosed with hypertension, the leading cause of cardiovascular disease and premature deaths in the world. Despite availability of effective drugs to control blood pressure, uncontrolled blood pressure and low adherence to antihypertensive drugs persist as major public health and clinical challenges. On average, 50% of adults adhere to chronic disease medications and lower levels of adherence are associated with worse blood pressure control and adverse outcomes. Many barriers to adherence are well known and have been targeted in interventions to improve medication adherence. As of yet, no single intervention has emerged as superior or even particularly effective in improving adherence. The investigators have recently identified unconscious, self-protective 'hidden motives' that contribute to nonadherence to chronic disease medications. There is a critical need to expand on this insight to test the potential for targeting individuals' 'hidden motives' for low adherence using an innovative learning process called Immunity-to-Change.

As a critical step in testing this intervention to target these 'hidden motives', the investigators will undertake a pilot study to assess the feasibility and acceptability of the Overcoming Immunity-to-Change intervention and determine effect sizes of the intervention on adherence, blood pressure (BP) control, and quality of life (QOL). The investigators will test the Immunity-to-Change intervention in a sample of nonadherent older adults with hypertension (n=18). Another sample of nonadherent older adults with hypertension will be monitored for comparison (n=18).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 55 and older, with the goal of a sex- and race-balanced sample
* Diagnosis of essential hypertension
* Uncontrolled hypertension
* Current treatment with antihypertensive medication
* Low antihypertensive pharmacy refill
* English speaking
* Telephone access
* Ability to read print on a computer screen and use the computer keyboard
* Written consent to participate and HIPAA authorization
* Written acceptance of study contract
* Approval of health care provider

Exclusion Criteria:

* Cognitive impairment
* Enrollment in another clinical trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence (PDC) | Baseline to 6 months
  Change in proportion of days covered (PDC) from baseline to 6 months

SECONDARY OUTCOMES:
Change in medication adherence (MMAS-8) | Baseline to 6 months
  Change in MMAS-8 score from baseline to 6 months
Change in medication adherence (KWood-4) | Baseline to 6 months
  Change in KWood-4 score from baseline to 6 months
Change in medication adherence (MMAS-8) | Baseline to 3 months
  Change in MMAS-8 score from baseline to 3 months
Change in medication adherence (KWood-4) | Baseline to 3 months
  Change in KWood-4 score from baseline to 3 months
Change in proportion with low adherence (PDC) | Baseline to 6 months
  Change in proportion with low adherence (PDC<0.8) from baseline to 6 months
Change in proportion with low adherence (MMAS-8) | Baseline to 6 months
  Change in proportion with low adherence (MMAS-8<6) from baseline to 6 months
Change in proportion with low adherence (KWood-4) | Baseline to 6 months
  Change in proportion with low adherence (KWood-4>0) from baseline to 6 months
Change in proportion with low adherence (MMAS-8) | Baseline to 3 months
  Change in proportion with low adherence (MMAS-8<6) from baseline to 3 months
Change in proportion with low adherence (KWood-4) | Baseline to 3 months
  Change in proportion with low adherence (KWood-4>0) from baseline to 3 months
Change in systolic blood pressure | Baseline to 6 months
  Change in systolic blood pressure from baseline to 6 months
Change in diastolic blood pressure | Baseline to 6 months
  Change in diastolic blood pressure from baseline to 6 months
Change in systolic blood pressure | Baseline to 3 months
  Change in systolic blood pressure from baseline to 3 months (if available from insurance records)
Change in diastolic blood pressure | Baseline to 3 months
  Change in diastolic blood pressure from baseline to 3 months (if available from insurance records)
Change in proportion with controlled blood pressure | Baseline to 6 months
  Change in proportion with controlled blood pressure (SBP<140 & DBP<90) from baseline to 6 months
Change in proportion with controlled blood pressure | Baseline to 3 months
  Change in proportion with controlled blood pressure (SBP<140 & DBP<90) from baseline to 3 months
Change in health-related quality of life | Baseline to 6 months
  Change in health-related quality of life score (SF-36) from baseline to 6 months
Change in health-related quality of life | Baseline to 3 months
  Change in health-related quality of life score (SF-36) from baseline to 3 months

OTHER OUTCOMES:
Change in hidden motives score | Baseline to 6 months
  Change in hidden motives score from baseline to 6 months
Change in hidden motives score | Baseline to 3 months
  Change in hidden motives score from baseline to 3 months
Change in explicit attitudes score | Baseline to 6 months
  Change in explicit attitudes score (Beliefs about Medicines Questionnaire) from baseline to 6 months
Change in explicit attitudes score | Baseline to 3 months
  Change in explicit attitudes score (Beliefs about Medicines Questionnaire) from baseline to 3 months
Change in implicit attitudes score | Baseline to 6 months
  Change in implicit attitudes score (d-score from single-category implicit association test) from baseline to 6 months
Change in explicit ambivalence score | Baseline to 6 months
  Change in explicit ambivalence score (absolute value of difference between standardized positive and negative explicit attitudes scores) from baseline to 6 months
Change in explicit ambivalence score | Baseline to 3 months
  Change in explicit ambivalence score (absolute value of difference between standardized positive and negative explicit attitudes scores) from baseline to 3 months
Change in implicit ambivalence score | Baseline to 6 months
  Change in implicit ambivalence score (absolute value of difference between standardized explicit and implicit attitude scores)
Change in short risk aversion switch point | Baseline to 6 months
  Change in short switch point on risk aversion scale from baseline to 6 months
Change in short risk aversion switch point | Baseline to 3 months
  Change in short switch point on risk aversion scale from baseline to 3 months
Change in long risk aversion switch point | Baseline to 6 months
  Change in long switch point on risk aversion scale from baseline to 6 months
Change in long risk aversion switch point | Baseline to 3 months
  Change in long switch point on risk aversion scale from baseline to 3 months
Change in risk valuation | Baseline to 6 months
  Change in value indicated on risk aversion scale from baseline to 6 months
Change in risk valuation | Baseline to 3 months
  Change in value indicated on risk aversion scale from baseline to 3 months
Change in medication-taking self-efficacy (MUSE) | Baseline to 6 months
  Change in score on MUSE medication-taking subscale from baseline to 6 months
Change in medication-taking self-efficacy (MUSE) | Baseline to 3 months
  Change in score on MUSE medication-taking subscale from baseline to 3 months
Change in learning-about-medications self-efficacy (MUSE) | Baseline to 6 months
  Change in score on MUSE learning-about-medications subscale from baseline to 6 months
Change in learning-about-medications self-efficacy (MUSE) | Baseline to 3 months
  Change in score on MUSE learning-about-medications subscale from baseline to 3 months
Change in self-efficacy (MUSE) | Baseline to 6 months
  Change in score on MUSE scale from baseline to 6 months
Change in self-efficacy (MUSE) | Baseline to 3 months
  Change in score on MUSE scale from baseline to 3 months
Change in self-efficacy (Self-Efficacy for Managing Chronic Disease) | Baseline to 6 months
  Change in score on SEMCD scale from baseline to 6 months
Change in self-efficacy (Self-Efficacy for Managing Chronic Disease) | Baseline to 3 months
  Change in score on SEMCD scale from baseline to 3 months
Change in chronic stress | Baseline to 6 months
  Change in chronic stress from baseline to 6 months, as measured by salivary cortisol
Change in perceived stress | Baseline to 6 months
  Change in score on 4-item version of Perceived Stress Scale from baseline to 6 months
Change in perceived stress | Baseline to 3 months
  Change in score on 4-item version of Perceived Stress Scale from baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Krousel-Wood, MD MSPH, Principal Investigator — Tulane University; Erin M Peacock, PhD MPH, Study Director — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krousel-Wood M, Kegan R, Whelton PK, Lahey LL. Immunity-to-change: are hidden motives underlying patient nonadherence to chronic disease medications? Am J Med Sci. 2014 Aug;348(2):121-8. doi: 10.1097/MAJ.0000000000000310. PMID 24978395